CLINICAL TRIAL: NCT02956330
Title: Retrospective Study of the Safety and Efficacy of Suprachoroidal CLS-TA in Combination With Intravitreal Aflibercept for the Treatment of Macular Edema Associated With RVO in Subjects Who Completed Parent Study CLS1003-201
Brief Title: Retrospective Study of the Safety and Efficacy of Patients With RVO in Subjects Who Completed Parent Study CLS1003-201
Status: Completed | Type: Observational
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLS1003-202
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: RVO; ME; Central Subfield Thickness; OCT; Optical Coherence Tomography; Cystoid Macular Edema; Subretinal Fluid; Eylea; Aflibercept; Anti-VEGF
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CLS1003-201: Those subjects whose parent study primary investigator has access to their medical records, following exit from CLS1003-201.

SUMMARY:
The purpose of this non interventional retrospective study is to continue to collect data from patients following their completion of Protocol CLS 1003-201: "Safety and Efficacy of Suprachoroidal CLS-TA with Intravitreal Aflibercept in Subjects with Macular Edema Following Retinal Vein Occlusion" (ie, the parent study).

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of up to 6 months for subjects that completed the parent study CLS1003-201. This study is designed to collect data from patients following their parent study exit visit, through either the time of the next treatment for RVO or at least 6 months following the parent study exit visit, whichever occurs first.

During this non-interventional retrospective study, the following data will be collected in an online questionnaire (or where required, on paper) provided by Clearside:

* Next RVO therapy administered (if applicable), including reason for treatment
* Continued documentation of current or changes in medical or ocular conditions following parent study
* Concomitant drug or therapy changes
* Visual acuity, including details on the method used in the assessment
* Central retinal thickness, including details on the equipment used in its determination
* Intraocular pressure, including details on the equipment used in its determination

Subjects will be selected based on parent study primary investigator's access to their medical records access, following exit from CLS1003-201. Data will also be collected on the total number of patients included in this non interventional study as well as reasons patients were excluded. Data will be summarized from the randomization treatment assignment in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Completed enrollment and did not receive additional aflibercept therapy in the Parent study, CLS1003-201

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately 30 adult subjects whose parent study primary investigator has access to their medical records, following exit from CLS1003-201.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Time to additional therapy for RVO | 6 months following exit from Parent study

SECONDARY OUTCOMES:
Mean change from baseline for intraocular pressure | 6 months following exit from Parent study
  Measured by applanation tonometry
Mean change from baseline in central subfield thickness | 6 months following exit from Parent study
  Based on spectral domain optical coherence tomography
Mean change from baseline in best corrected visual acuity | 6 months following exit from Parent study
  Based on ETDRS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (1):
- San Antonio, Texas, United States